CLINICAL TRIAL: NCT00006157
Title: Multicenter Trial of Functional Bowel Disorders
Brief Title: Treatment of Functional Bowel Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: FBD (completed); R01DK049334 (NIH)
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Irritable Bowel Syndrome; Constipation; Abdominal Pain; Functional Colonic Diseases
Keywords: Functional bowel disorder; Irritable bowel syndrome; Painful constipation; Unspecified functional bowel disorder; Chronic functional abdominal pain; Cognitive-behavioral psychological treatment; IBS; CFAP
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation; Abdominal Pain; Colonic Diseases, Functional | interventions — Desipramine

INTERVENTIONS:
Drug: Desipramine
Behavioral: Cognitive Behavioral Treatment

SUMMARY:
The primary purpose for this study is to compare clinical treatments for patients with functional bowel disorders (irritable bowel syndrome, abdominal pain, painful constipation) in women. We also plan to: 1) determine what clinical features (medical or psychological) determine which patients will improve to these treatments, and 2) understand if there are any physiological features that relate to improvement in symptoms and response to the treatments.

We will compare a psychological treatment (cognitive-behavioral therapy - CBT) with education/attention placebo, and an antidepressant drug (desipramine) with a pill placebo. This is the first large-scale study designed to determine the therapeutic effects of these methods, and to also determine interactions among physiologic measures, psychologic and sociodemographic factors, severity of symptoms, and therapeutic improvement including quality of life.

DETAILED DESCRIPTION:
Female patients (aged 18-65) with FBD (irritable bowel syndrome, painful constipation and/or functional abdominal pain) will be enrolled at UNC-Chapel Hill and Toronto, Canada. A severity index will determine recruitment into the group of moderate FBD (200 patients) and severe FBD (100 patients). Each group will be randomized into the three treatment arms (cognitive-behavioral treatment, desipramine, and education/attention placebo), treated over a 12-week period, and followed for one year. Outcome measures will include symptoms (standardized abdominal pain, stool form and frequency) using diary cards, daily functional status (Sickness Impact Profile), depression (HAM-D) and psychological distress (SCL-90), physiological measures (enhanced rectal motility and visceral sensation), and health care use. Multivariate statistical methods with a hierarchical design will be applied to the data to assure maintenance of statistical power over multiple tests of overlapping groups.

The results of this study should significantly improve our understanding of this complicated syndrome that lowers the quality of life and economic productivity of large numbers of women. The clinical impact of the study, in providing physicians with scientific evidence of the efficacy of treatments of FBD that are commonly used in practice, is significant. We anticipate that this study will provide clinicians with predictors of success among types of FBD patients and types of therapy that will improve symptoms and quality of life, and reduce the health care costs associated with this common syndrome while improving patient-physician satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Literate, female patients aged 18-65.
* Symptoms present at least 2 days/week for greater than 6 months.
* Diagnosis of functional bowel disorder (to be subcategorized using ''Rome'' Criteria.
* Moderate (MFBD) or severe (SFBD) functional bowel disorder (FBD) based on the Functional Bowel Disorder Severity Index (FBDSI) developed in our pilot study. SFBD will be defined as a score of 110 and MFBD will be defined as a score between 36 and 110.
* Discontinuation of all antidepressant medications for at least 3 months.
* Use of acceptable method of birth control.

Exclusion Criteria:

* Evidence of lactose intolerance to explain bowel symptoms.
* Heart disease.
* Cardiac arrhythmias.
* Severe psychiatric disorder (e.g., bipolar, suicide attempts).
* Previous use of desipramine.
* Glaucoma.
* Urinary retention.
* Pregnancy.
* Alcohol consumption 3oz/day that would preclude participation or prevent data assessment.
* Systemic gastrointestinal diseases or previous surgery that would interfere with the interpretation of symptoms or physiology.
* Bipolar disorder.
* Schizophrenia.
* Substance abuse/dependency.
* Previous use of desipramine.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1996-07; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Overall Officials: Douglas A. Drossman, M.D., Principal Investigator — Univ of North Carolina at Chapel Hill; William E. Whitehead, PhD, Study Chair — Univ of North Carolina at Chapel Hill; Brenda Toner, PhD, Study Chair — Centre for Addiction and Mental Health, Clark Site; Nick Diamant, MD, Study Chair — The Toronto Western Hospital
Locations (2):
- UNC Center for Functional GI Motility Disorders, Chapel Hill, North Carolina, United States
- Centre for Addiction and Mental Health, Clark Site, Toronto, Ontario, Canada

REFERENCES:
- See also: The website for the UNC Center for Functional GI and Motility Disorders contains information on our center, functional bowel disorders, current clinical trials, and other FBD resources. — http://www.med.unc.edu/ibs